CLINICAL TRIAL: NCT00576654
Title: A Phase I Dose-Escalation Study of Oral ABT-888 (NSC #737664) Plus Intravenous Irinotecan (CPT-11, NSC#616348) Administered in Patients With Advanced Solid Tumors
Brief Title: Veliparib and Irinotecan Hydrochloride in Treating Patients With Cancer That Is Metastatic or Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-01057; NCI-2009-01057 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1410014852; CDR0000579642; HIC 1410014852; 2007-014; HIC1410014852; 7977 (Other: Yale University Cancer Center LAO); 7977 (Other: CTEP); R21CA135572 (NIH); U01CA062487 (NIH); U01CA062490 (NIH); UM1CA186689 (NIH); UM1CA186709 (NIH)
Record Dates: First submitted 2007-12-18; First posted 2007-12-19 (Estimated); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Advanced Malignant Solid Neoplasm; Metastatic Malignant Solid Neoplasm; Triple-Negative Breast Carcinoma; Unresectable Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis; Triple Negative Breast Neoplasms | interventions — Irinotecan; veliparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dose escalation (irinotecan hydrochloride and veliparib) (Experimental): Patients receive irinotecan hydrochloride IV over 90 minutes on days 1 and 8 and veliparib PO BID on days -1 to 14 (days 3-14 of course 1 only). Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Irinotecan Hydrochloride; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Veliparib
- Expansion portion (irinotecan hydrochloride and veliparib) (Experimental): Patients receive irinotecan hydrochloride IV over 90 minutes on days 1 and 8 and veliparib PO BID on days 1-15 (days 2-15 of course 1 only). Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Irinotecan Hydrochloride; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Veliparib
- Intermittent dose escalation (irinotecan, ABT-888) (Experimental): Patients receive irinotecan hydrochloride IV over 90 minutes on days 3 and 10 and veliparib PO BID on days 1 to 4 and 8-11. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Irinotecan Hydrochloride; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Veliparib

INTERVENTIONS:
Drug: Irinotecan Hydrochloride — Given IV
  Other Names: Campto; Camptosar; Camptothecin 11; Camptothecin-11; CPT 11; CPT-11; CPT11; Irinomedac; Irinotecan Hydrochloride Trihydrate; Irinotecan Monohydrochloride Trihydrate; U 101440E; U-101440E; U101440E
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Veliparib — Given PO
  Other Names: ABT 888; ABT-888; ABT888; PARP-1 inhibitor ABT-888

SUMMARY:
This phase I trial studies the side effects and best dose of veliparib when given together with irinotecan hydrochloride in treating patients with cancer that has spread to other parts of the body or that cannot be removed by surgery. Irinotecan hydrochloride can kill cancer cells by damaging the deoxyribonucleic acid (DNA) that is needed for cancer cell survival and growth. Veliparib may block proteins that repair the damaged DNA and may help irinotecan hydrochloride to kill more tumor cells. Giving irinotecan hydrochloride together with veliparib may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the optimal biologic dose (OBD) for poly (adenosine diphosphate [ADP]-ribose) polymerase (PARP) inhibition using irinotecan (irinotecan hydrochloride) (once weekly intravenously in 2 of 3 weeks), in combination with ABT-888 (veliparib) (twice daily orally for 2 of 3 weeks). (ORIGINAL DOSE ESCALATION PORTION) II. To determine the recommended phase II dose (RP2D) for irinotecan (once weekly intravenously in 2 of 3 weeks), in combination with ABT-888 (twice daily orally for 2 of 3 weeks), determined by evaluating the feasibility, safety, dose limiting toxicities and the maximally tolerated dose. (ORIGINAL DOSE ESCALATION PORTION) III. To determine the safety profile of irinotecan in combination with ABT-888: the incidence of adverse events (AEs) and clinically significant changes in laboratory tests, electrocardiograms (ECGs), and vital signs. (ORIGINAL DOSE ESCALATION PORTION) IV. To determine the safety profile of irinotecan in combination with ABT-888 at the recommended phase II dose: the incidence of adverse events (AEs) and clinically significant changes in laboratory tests, ECGs, and vital signs. (ORIGINAL DOSE ESCALATION PORTION) V. To determine the recommended phase II dose (RP2D) of each drug for irinotecan (once weekly intravenously in 2 of 3 weeks), in combination with ABT-888 (twice daily orally for intermittent dosing days 1 to 4 and days 8 to 11 of each cycle), determined by evaluating the feasibility, safety, dose limiting toxicities and the maximally tolerated dose (MTD). (DOSE ESCALATION FOR INTERMITTENT ABT-888 PORTION) VI. To determine the safety profile of irinotecan in combination with ABT-888: the incidence of adverse events (AEs) and clinically significant changes in laboratory tests, and vital signs. (DOSE ESCALATION FOR INTERMITTENT ABT-888 PORTION) VII. To determine the safety profile of irinotecan in combination with ABT-888 at the recommended phase II dose: the incidence of adverse events (AEs) and clinically significant changes in laboratory tests, and vital signs. (DOSE ESCALATION FOR INTERMITTENT ABT-888 PORTION)

SECONDARY OBJECTIVES:

I. To determine the pharmacokinetic (PK) profile of ABT-888. II. To determine the PK profile of irinotecan (CPT-11) both as a single agent and in combination with ABT-888.

III. To determine the tumor response as assessed by the Response Evaluation Criteria in Solid Tumors (RECIST).

IV. To determine the tumor response as assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). (DOSE ESCALATION FOR INTERMITTENT ABT-888 PORTION) V. To describe response rate (RR) in patients. (DOSE ESCALATION FOR INTERMITTENT ABT-888 PORTION)

TERTIARY OBJECTIVES:

I. Pharmacodynamic (PD) biomarker response: PARP inhibition in peripheral blood mononuclear cells (PBMC) by measurement of PAR levels. (ORIGINAL DOSE ESCALATION PORTION) II. DNA damaging effects of irinotecan and the combination of irinotecan with ABT-888: levels of gamma H2A histone family, member X (gamma-H2AX) and RAD51 recombinase (Rad51) formation in tumor tissue. (ORIGINAL DOSE ESCALATION PORTION) III. Relevance of cytochrome P450 family 2, subfamily C, polypeptide 9 (CYP2C9) and 2C19 polymorphisms, uridine 5'-diphosphosphate (UDP) glucuronosyltransferase 1 family, polypeptide A1 (UGT1A1) polymorphism, and ATP-binding cassette, sub-family G (WHITE), member 2 (ABCG2) polymorphism to the pharmacokinetics of irinotecan and/or ABT-888. (ORIGINAL DOSE ESCALATION PORTION) IV. To explore whether a positive gamma-H2AX response in tumor tissue at 4-6 hours (hrs) is reflected in circulating tumor cells (CTCs) between 8-24 hrs but not at 4-6 hrs, as predicted. (EXPANSION PORTION) V. To explore whether PARP inhibition increases gamma-H2AX response of CTCs to plasma drug by 4-6 hrs after CPT-11 administration. (EXPANSION PORTION) VI. To explore whether PARP inhibition increases gamma-H2AX response of tumor cells to tissue drug level, as indicated by CTCs at 8-24 hrs after CPT-11. (EXPANSION PORTION) VII. To explore when the gamma-H2AX response peak in CTCs occurs, indicating a response in tumor. (EXPANSION PORTION) VIII. To explore whether there is a tumor switch between gamma-H2AX and excision repair cross-complementation group 1 (ERCC1)-mediated repair in the presence of PARP inhibition, (i.e., repeat initial PBMC and tumor findings). (EXPANSION PORTION) IX. To perform analysis of CTCs at day 15 to help guide alteration in ABT-888 drug administration schedule (continuous administration). (EXPANSION PORTION) X. To sequence the genome and transcriptome from both normal and tumor tissue from each study patient in the expansion cohort to evaluate point mutations, structural changes and copy number events. (EXPANSION PORTION) XI. To evaluate the damaging effects of irinotecan and the combination of irinotecan with ABT-888 by examining levels of Rad51 formation in tumors. (EXPANSION PORTION) XII. To evaluate the percentage of breast cancer stem cells (BCSC) in serial breast tumor biopsies before and after irinotecan alone and after 1 cycle of treatment with the combination of irinotecan and ABT-888. (EXPANSION PORTION) XIII. To perform molecular profiling of the tumor cell and BCSC populations before and after irinotecan alone and after 1 cycle of treatment with the combination of irinotecan and ABT-888. (EXPANSION PORTION) XIV. To compare Rad51 foci in aldehyde dehydrogenase-positive (ALDH+) stem cell populations to the bulk tumor cells. (EXPANSION PORTION) XV. To develop assays to detect trapping of PARP1 and 2 in tumor biopsy tissue in response to treatment with irinotecan plus a PARP inhibitor, in this case ABT-888. (DOSE ESCALATION FOR INTERMITTENT ABT-888 PORTION) XVI. Additional exploratory assay to be named later. (DOSE ESCALATION FOR INTERMITTENT ABT-888 PORTION)

OUTLINE: This is a dose-escalation study of veliparib. Patients are assigned to 1 of 3 cohorts.

DOSE ESCALATION: Patients receive irinotecan hydrochloride intravenously (IV) over 90 minutes on days 1 and 8 and veliparib orally (PO) twice daily (BID) on days -1 to 14 (days 3-14 of course 1 only). Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

EXPANSION PORTION: Patients receive irinotecan hydrochloride IV over 90 minutes on days 1 and 8 and veliparib PO BID on days 1-15 (days 2-15 of course 1 only). Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

INTERMITTENT DOSE ESCALATION: Patients receive irinotecan hydrochloride IV over 90 minutes on days 3 and 10 and veliparib PO BID on days 1 to 4 and 8-11. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed diagnosis of malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective or for whom CPT-11 treatment would be a viable therapy regimen; patients with solid hematologic malignancies (Hodgkin's and non-Hodgkin's lymphomas) may be included as long as a bone marrow has been performed within 6 weeks of treatment
* Patients enrolled on the expansion portion of the study will consist of two cohorts: those patients who are triple-negative, BRCA-mutant positive and those patients who have triple-negative, non-BRCA mutated breast cancer
* Patients enrolled on the dose escalation for intermittent ABT-888 portion of the study must histologically or cytologically confirmed diagnosis of malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective or for whom CPT-11 treatment would be a viable therapy regimen; patients with solid hematologic malignancies (Hodgkin's and non-Hodgkin's lymphomas) may be included as long as a bone marrow has been performed within 6 weeks of treatment
* Patient must have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) guidelines
* Patients must have tumors determined to be easily accessible for biopsy (e.g. pleural-based lesions, peripheral lymph nodes, soft tissue metastases, large liver metastases, etc)
* Prior chemotherapy is allowed; patients must not have received chemotherapy for 4 weeks prior to the initiation of study treatment and must have full recovery from any acute effects of any prior chemotherapy; patients must not have had nitrosoureas or mitomycin C for 6 weeks prior to the initiation of study treatment
* Prior radiation therapy is allowed; patients must not have received minimal radiation therapy (=< 5% of their total marrow volume) within 3 weeks prior to the initiation of study treatment; otherwise, patients must not have received radiation therapy (> 5% of their total marrow volume) within 4 weeks prior to the initiation of study treatment; patients who have received prior radiation to 50% or more of their total marrow volume will be excluded
* Prior experimental (non-Food and Drug Administration [FDA] approved) therapies and immunotherapies are allowed; patients must not have received these therapies for 4 weeks prior to the initiation of study treatment and must have full recovery from any acute effects of these therapies
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 12 weeks
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelets (PLT) >= 100,000/mcL
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x upper limit of normal (ULN); if liver metastases are present, =< 5 x ULN
* Bilirubin =< 1.5 x ULN
* Creatinine =< 1.5 x ULN OR calculated or measured creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine above institutional normal
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for three months following completion of study therapy; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document
* All patients must provide archival tissue block or paraffin sample from archival tissue block (approximately 10 sections) for use in pharmacodynamic correlative studies (NOT required for patients enrolled on the dose escalation for intermittent ABT-888 portion of the study)

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier; patients who have been administered ABT-888 as part of a single or limited dosing study, such as a phase 0 study, should not necessarily be excluded from participating in this study solely because of receiving prior ABT-888
* Patients may not have received any other investigational agents within 4 weeks of study entry
* History of allergic reactions attributed to the following:

  * Camptothecin derivatives (e.g., topotecan [topotecan hydrochloride], irinotecan, or exatecan [exatecan mesylate])
  * Any ingredients contained within the liquid irinotecan solution (e.g., sorbitol) or
  * Any antiemetics or antidiarrheals appropriate for administration with study therapy (e.g., loperamide or dexamethasone)
* Patients must not receive any other anti-cancer therapy (cytotoxic, biologic, radiation, or hormonal other than for replacement) while on this study except for medications that are prescribed for supportive care but may potentially have an anti-cancer effect (i.e. megestrol acetate, bisphosphonates); these medications must have been started 1 month prior to enrollment on this study; in addition, men receiving treatment for prostate cancer will be maintained at castrate levels of testosterone by continuation of luteinizing-releasing hormone agonists
* Patients with uncontrolled seizures
* Patients with known active brain metastases should be excluded from this clinical trial; patients with prior treated brain metastases are allowed, providing that they were not accompanied by seizures and that a baseline brain magnetic resonance imaging (MRI) scan prior to study entry demonstrates no current evidence of brain metastases; all patients with central nervous system (CNS) metastases must be stable for > 3 months after treatment and off steroid treatment prior to study enrollment
* Any patient requiring chronic maintenance of white blood cell counts or granulocyte counts through the use of growth factor support (e.g. Neulasta, Neupogen)
* Any patient requiring cytochrome P450 family 3, subfamily A, polypeptide 4 (CYP3A4) isoform-inducing drugs (e.g. phenytoin, phenobarbital, carbamazepine, rifampin, rifabutin, ketoconazole, St. John's wort) will be excluded; CYP3A4-inducing drugs should be discontinued at least 2 weeks prior to the first cycle of irinotecan
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia or
  * Psychiatric illness or social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with ABT-888
* Patients who are unable to reliably tolerate and/or receive oral medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2008-03-18 (Actual); Primary Completion 2020-01-16 (Actual); Study Completion 2020-01-16 (Actual)

PRIMARY OUTCOMES:
Optimal biologic dose (OBD) | Up to day 9 of course 1
  Defined as the dose level at which no greater inhibition of poly(ADP-ribose) (PAR) levels in tumor cells is identified, relative to the next lower dose.
Maximum administered dose of study drugs | Up to 21 days
  Defined as the dose level at which at least 2 of 6 patients develop dose-limiting toxicity (DLT) as graded by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Maximally tolerated dose (MTD) of study drugs | Up to 21 days
  Defined as the dose at which no more than 1 patient of 6 develops DLT as graded by the NCI CTCAE version 5.0.
Recommended phase II dose (RP2D) of study drugs | Up to 21 days
  Defined as the MTD if DLTs are observed before achieving the OBD, or the OBD if DLTs are not observed before reaching the OBD as graded by the NCI CTCAE version 5.0.

SECONDARY OUTCOMES:
Incidence of adverse events (AEs), graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 | Up to 30 days
  Described by point estimates and exact 90% confidence intervals.
Tumor response | Up to 30 days
  Evaluated using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

OTHER OUTCOMES:
Change in poly(ADP-ribose) polymerase (PARP) levels in peripheral blood mononuclear cells (PBMCs) | Baseline to up to 10 days
  Summarized with standard descriptive statistics (N, median, mean, standard deviation, minimum, maximum, and 90% confidence interval for the mean).
Pharmacokinetic (PK) profile of veliparib | Baseline and at days 1, 2, and 3 of course 1 and days 1, 8, 9, and 10 of course 2
  Summarized with standard descriptive statistics (N, median, mean, standard deviation, minimum, maximum, and 90% confidence interval for the mean).
Poly(ADP-ribose) (PAR) activity inhibition in peripheral blood mononuclear cells and tumor cells | Up to 10 days
  Will be measured.
Change in gamma-H2AX foci and/or Rad51 levels | Baseline to up to day 9 of course 1
  Summarized with standard descriptive statistics (N, median, mean, standard deviation, minimum, maximum, and 90% confidence interval for the mean).
Pharmacodynamic (PD) parameters | Up to 30 days
  Will be summarized descriptively, by dose level and overall and will be summarized with standard statistics (N, median, mean, standard deviation, minimum, maximum, and 90% confidence interval for the mean).
Pharmacokinetic (PK) parameters of irinotecan hydrochloride | Baseline, 5.5 hours after infusion, and 28 hours after infusion of day one of course 1
  Will be summarized descriptively within each cytochrome p450, family 2, subfamily C, polypeptide 9 (CYP2C9) polymorphism category, by dose level and overall.
Circulating tumor cell (CTC) counts | Up to day 15
  Will be measured.
Excision repair cross-complementation group 1 (ERCC1) expression levels | Up to day 8
  Will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia M LoRusso, Principal Investigator — Yale University Cancer Center LAO
Locations (5):
- United States (5):
  - Yale University, New Haven, Connecticut
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Covenant Medical Center Harrison, Saginaw, Michigan